CLINICAL TRIAL: NCT04958954
Title: Post-Marketing Safety of SARS-CoV-2 mRNA-1273 Vaccine in the US: Active Surveillance, Signal Refinement and Self-Controlled Risk Interval (SCRI) Signal Evaluation in HealthVerity
Brief Title: Post-Marketing Safety Study of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) mRNA-1273 COVID-19 Vaccine in the United States
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P903; EUPAS41392 (Other: EU PAS Register Number)
Record Dates: First submitted 2021-07-09; First posted 2021-07-12 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (4):
- Cohort 1a: Pre-COVID: All participants meeting eligibility criteria in the Pre-COVID-19 period (immediately preceding the emergence of COVID-19) (Time Period 1) from 01 December 2018 to 30 November 2019
- Cohort 1b: Pre-COVID: All participants with evidence of an influenza vaccination and meeting eligibility criteria in the Pre-COVID-19 period (immediately preceding the emergence of COVID-19) (Time Period 1) from 01 December 2018 to 30 November 2019
- Cohort 2: Active-COVID: All participants meeting eligibility criteria in the Active-COVID-19 period, Pre-Emergency Use Authorization (EUA) period (following the emergence of COVID-19 but before the first COVID-19 vaccine EUA) (Time Period 2) from 01 December 2019 to 10 December 2020 (1 day prior to first United States SARS-CoV-2 vaccine EUA)
- Cohort 3: Post-EUA: All mRNA-1273 vaccinated participants meeting eligibility criteria in the Post-EUA period (Time Period 3) from date of first United States SARS-CoV-2 vaccine EUA to 31 December 2022

SUMMARY:
The goal of this study is to add to the ongoing active and passive safety signal detection through signal refinement and, if needed, evaluation of potential safety signals related to taking the SARS-CoV-2 mRNA-1273 vaccine.

DETAILED DESCRIPTION:
This retrospective observational cohort study will use secondary, de-identified individual-level medical and pharmacy claims data provided by HealthVerity.

ELIGIBILITY:
Inclusion Criteria:

* Included in a health plan covered by HealthVerity database
* Covered by a health plan during at least 1 period of interest (pre-COVID-19, active-COVID-19, and post-EUA periods), but not necessarily the full period.
* Demonstrate an AESI specified clean period of continuous baseline enrollment or activity before the period of interest (pre-COVID-19, active-COVID-19, and post-EUA periods) during which the participant is covered.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from HealthVerity's aggregated medical and pharmacy claims database that represents healthcare utilization for over 140 million participants between 01 December 2017 and the end of the study period (31 December 2022).
Sampling Method: Non-Probability Sample
Enrollment: 50000000 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events of Special Interests (AESIs) | Index date (that is, first day of health plan eligibility within the applicable time period where all study entry criteria are met) through end of data availability or earliest event (maximum of 751 days depending on duration of capture in the database)

CONTACTS AND LOCATIONS:
Locations (1):
- Aetion Inc., New York, New York, United States